CLINICAL TRIAL: NCT05774431
Title: Disparities in the Proportion of Ticagrelor and Prasugrel-eligible Patients with Acute Coronary Syndrome in a Real-world Registry
Acronym: AZ-DAPT
Status: Completed | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Mustafa Yildirim, Principal Investigator, University Hospital Heidelberg
Other Study IDs: AZ-DAPT
Record Dates: First submitted 2023-03-06; First posted 2023-03-17 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: There was no intervention necessary. — There was no intervention necessary.

SUMMARY:
The primary objective of this study is to compare patients eligible for ASS and Ticagrelor against those eligible for ASS and Prasugrel. The available information regarding relative and absolute exclusion criteria outlines reasons for disqualification from either drug.

The secondary objectives of the study are to:

* Assess the proportion of patients who received ASS and Ticagrelor in the study cohort.
* Compare the proportion of patients who received ASS and Ticagrelor against the proportion of patients who qualify for DAPT with ASS and Ticagrelor (eligible group).
* Describe the antithrombotic treatment, including antiplatelet monotherapies, and antiplatelet therapies with or without anticoagulation.

The investigators will use these objectives to evaluate the effectiveness and appropriateness of the different antiplatelet therapies in the study population. Participants will not be personally identified in any reports or publications resulting from this study.

DETAILED DESCRIPTION:
This retrospective single-center study at University Hospital of Heidelberg aims to consecutively screen all patients with suspected ACS over a 24-month period. Patients will be managed in a chest pain unit (CPU), which is a specialized ED led by a cardiologist and requires certification by the German Cardiac Society (Deutsche Gesellschaft für Kardiologie; DGK). More than 320 certified CPUs are distributed across Germany and represent the preferred facilities for evaluating patients with suspected ACS. CPU organization and certification requirements have been previously published.

The ED is under the supervision of a senior cardiologist who is responsible for decisions regarding admission or discharge, selection of antiplatelet and antithrombotic drugs, and indication and timing of an invasive strategy. All patients will undergo a clinical assessment, including medical history, physical examination, 12-lead ECG, continuous ECG monitoring, pulse oximetry, and standard blood tests. The standard 12-lead ECG includes routinely precordial leads V7-V9. Results will be reported on the electronic patient record and communicated to the clinicians responsible for patient care.

There is unlimited access to coronary angiography or other diagnostic resources as per the required criteria for certification of a CPU. Although STEMI patients were not excluded from the analysis, patients with qualifying ST-segment elevations or a presumably new bundle branch block were primarily seen in the catheterization laboratory bypassing the ED. All decisions for adjunctive pharmacological treatments are left to the discretion of the invasive cardiologist before transfer back for observation to the coronary care ward or to the ED.

Acute myocardial infarction (MI) will be diagnosed in-hospital by treating clinicians based on all clinical information, using the diagnostic criteria of the 3rd or 4th universal MI definition. For research purposes, two cardiologists will retrospectively confirm ED diagnoses, with a third cardiologist consulted in case of discordance. All files of patients with confirmed ACS will be screened for information on body weight, pretreatment with P2Y12-Inhibitors before hospital admission, pre-treatment with oral anticoagulants before index admission, or new requirement for oral anticoagulation. Data on age, selection of antiplatelet drugs, invasive strategy including rates of coronary angiography, PCI, CABG, a planned conservative, or conservative therapy in the case of complex coronary angiography or failed PCI were already collected in the electronic registry database, and findings from this registry have been previously published.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Clinical symptoms of acute coronary syndrome

Exclusion Criteria:

* hemodialysis
* Atrial tachycardia with accompanying symptoms, but without clinical suspicion of an ACS (Acute Coronary Syndrome).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this retrospective single center study, we will consecutively screen all patients with suspected acute coronary syndrome presenting to the Chest Pain Unit (CPU) of the University Hospital of Heidelberg between 1st of July 2016 and 30th of June 2018. Patients will be managed in CPU, which represents a specialized emergency department (ED) that is led by a cardiologist and requires certification by the German Cardiac Society (Deutsche Gesellschaft für Kardiologie; DGK).
Sampling Method: Probability Sample
Enrollment: 6789 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Comparison of Eligible Patients for Dual Antiplatelet Therapy: ASS and Ticagrelor vs ASS and Prasugrel | 24 months
  Comparing patients who are eligible for ASS and Ticagrelor against those who are eligible for ASS and Prasugrel

SECONDARY OUTCOMES:
Proportion of Patients Receiving ASS and Ticagrelor: Comparison to Eligible Group and Description of Antithrombotic Treatment in Study Cohort | 24 months
  Assessing the proportion of patients who received ASS and Ticagrelor in the study cohort, to compare the proportion of patients who received ASS and Ticagrelor against the proportion of patients who qualify for DAPT with ASS and Ticagrelor (eligible group) and to describe the antithrombotic treatment, i.e. antiplatelet monotherapies, antiplatelet therapies with or without anticoagulation.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yildirim M, Reich C, Salbach C, Biener M, Mueller-Hennessen M, Sorensen NA, Haller PM, Blankenberg S, Neumann JT, Twerenbold R, Frey N, Giannitsis E. Identification of patients with suspected NSTE-ACS in the observe zone: evaluating GRACE 1.0 score and a biomarker panel for risk stratification and management optimization. Clin Res Cardiol. 2025 Jun;114(6):783-795. doi: 10.1007/s00392-025-02642-3. Epub 2025 Apr 14. PMID 40227426
- [Derived] Yildirim M, Mueller-Hennessen M, Milles BR, Biener M, Hund H, Frey N, Giannitsis E, Salbach C. Real-World Evidence on Disparities on the Initiation of Ticagrelor Versus Prasugrel in Patients With Acute Coronary Syndrome. J Am Heart Assoc. 2023 Aug 15;12(16):e030879. doi: 10.1161/JAHA.123.030879. Epub 2023 Aug 10. PMID 37581388